CLINICAL TRIAL: NCT00355706
Title: Effectiveness of Thoracic Facet Joint Nerve Blocks: A Randomized, Prospective, Double-Blind Controlled Evaluation
Brief Title: Effectiveness of Thoracic Facet Joint Nerve Blocks
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pain Management Center of Paducah (Other)
Responsible Party: Principal Investigator, Laxmaiah Manchikanti, MD, Medical Director, Pain Management Center of Paducah
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: protocol 5
Record Dates: First submitted 2006-07-24; First posted 2006-07-25 (Estimated); Results first posted 2013-11-26 (Estimated); Last update posted 2020-03-10 (Actual); Status verified 2020-03

CONDITIONS: Low Back Pain
Keywords: chronic low back pain; thoracic facet joint; nerve block
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group I - without Steroids (Active Comparator): Thoracic Facet Joint Nerve Blocks with Local Anesthetic(0.25% Bupivacaine)
  Interventions: Procedure: Thoracic facet joint nerve blocks
- Group II - with steroid (Active Comparator): Thoracic Facet Joint Nerve Blocks with Local Anesthetic (0.25% Bupivacaine) and Sterioids(0.15 mg of non-particulate betamethasone)
  Interventions: Procedure: Thoracic facet joint nerve blocks

INTERVENTIONS:
Procedure: Thoracic facet joint nerve blocks — Thoracic medial branch blocks
  Other Names: Thoracic medial branch blocks

SUMMARY:
1. To demonstrate whether:

   i. Facet joint nerve blocks have therapeutic value beyond the duration of local anesthetic effect.

   ii. Addition of Depo-steroid provides additional relief of thoracic facet joint pain when used with facet joint nerve blocks.
2. To demonstrate whether or not there are clinically significant improvements in function of patients who receive thoracic facet joint nerve block with Depo-steroid compared to patients randomized to Group I who receive only local anesthetic blocks.
3. To determine the adverse event profile in both groups

DETAILED DESCRIPTION:
Participants Study participants were recruited at the interventional pain management practice from consecutive new patients presenting with thoracic pain. One hundred patients were included and randomly assigned to one of 2 groups; either a local anesthetic only group (Group I) or a local anesthetic with steroid group (Group II), with 50 patients in each group. Patients meeting the inclusion criteria were eligible to undergo diagnostic thoracic facet joint nerve blocks. Only patients positive for controlled comparative local anesthetic blocks met the criteria for inclusion for thoracic medial branch blocks.

Inclusion and Exclusion Criteria Only patients with nonspecific mid-back or upper back pain without suspected disc herniation, radiculitis, thoracic fracture, stenosis, or intercostal neuritis were included. Further, patients suspected of disc-related pain with radicular symptoms were also excluded, based on radiologic testing and symptomatology involving radicular or chest wall pain. Patients also should have previously received conservative management with physical therapy, chiropractic manipulation exercises, drug therapy, and bed rest, and so forth, but continued to have pain.

Further inclusion criteria were a diagnosis of thoracic facet joint pain by means of controlled comparative local anesthetic blocks; patients who were over 18 years of age; patients with a history of chronic function-limiting mid-back or upper back pain of at least 6 months duration; and patients who where competent to understand the study protocol and provide voluntary, written informed consent, and participate in the outcome measurements. A negative or false-positive response to controlled comparative local anesthetic blocks, uncontrollable to heavy opioid use (morphine equivalent of 300 mg), uncontrolled

ELIGIBILITY:
Inclusion Criteria:

Positive for facet joint pain with comparative local anesthetic blocks

Candidates are over 18 years of age

Subjects with a history of chronic, function limiting neck pain of at least six months in duration Subjects who are able to give voluntary, written informed consent to participate in this investigation Subjects who, in the opinion of the Investigator, are able to understand this investigation, co-operate with the investigational procedures and are willing to return to the center for all the required post-operative follow-ups The subject has not had recent surgical procedures within the last three months.

-

Exclusion Criteria:

* Negative or false-positive response to controlled comparative local anesthetic blocks

Narcotic use of greater than Hydrocodone 100 mg/day, Methadone 80 mg or Morphine 100 mg, or dose equivalent

Uncontrolled major Depression or uncontrolled psychiatric disorders

Uncontrolled or acute medical illnesses including coagulopathy, renal insufficiency, chronic liver dysfunction, progressive neurological deficit, urinary sphincter dysfunction, infection, increased intercranial pressure, pseudotumor cerebri, intercranial tumors, unstable angina, and severe chronic obstructive pulmonary disease.

Chronic severe conditions that could interfere with the interpretations of the outcome assessments for pain and bodily function

Women who are pregnant or lactating

Subjects who have participated in a clinical study with an investigational product within 30 days of enrollment

Patients with multiple complaints involving concomitant hip osteoarthritis, will not be amenable to study due to the overlap of pain complaints.

Inability to achieve appropriate positioning and inability to understand informed consent and protocol History of adverse reaction to local anesthetic or anti-inflammatory drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2003-08; Primary Completion 2006-07 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Laxmaiah Manchikanti, MD, Principal Investigator — Ambulatory Surgery Center
Locations (1):
- Ambulatory Surgery Center, Paducah, Kentucky, United States

REFERENCES:
- [Result] Manchikanti L, Singh V, Falco FJ, Cash KA, Pampati V, Fellows B. The role of thoracic medial branch blocks in managing chronic mid and upper back pain: a randomized, double-blind, active-control trial with a 2-year followup. Anesthesiol Res Pract. 2012;2012:585806. doi: 10.1155/2012/585806. Epub 2012 Jul 19. PMID 22851967
- [Derived] Manchikanti L, Singh V, Falco FJ, Cash KA, Pampati V, Fellows B. Comparative effectiveness of a one-year follow-up of thoracic medial branch blocks in management of chronic thoracic pain: a randomized, double-blind active controlled trial. Pain Physician. 2010 Nov-Dec;13(6):535-48. PMID 21102966
- [Derived] Manchikanti L, Singh V, Falco FJ, Cash KA, Pampati V. Effectiveness of thoracic medial branch blocks in managing chronic pain: a preliminary report of a randomized, double-blind controlled trial. Pain Physician. 2008 Jul-Aug;11(4):491-504. PMID 18690278
- See also: The Role of Thoracic Medial Branch Blocks in Managing Chronic Mid and Upper Back Pain: A Randomized, Double-Blind, Active-Control Trial with a 2-Year Followup — http://www.ncbi.nlm.nih.gov/pmc/articles/PMC3407605/pdf/ARP2012-585806.pdf

RESULTS

PARTICIPANT FLOW:
Groups:
- Group I - Without Steroids: Group I - Thoracic medial branch blocks with local anesthetics
- Group II - With Steroids: Group II - Thoracic medial branch blocks with bupivacaine and steroid
Period: Overall Study
Arm/Group | Group I - Without Steroids | Group II - With Steroids
Started | 50 | 50
Completed | 50 | 50
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Group I - With Local Anesthetics: Group I - Thoracic medial branch blocks with local anesthetics
- Group II - With Bupivacaine and Steroid: Group II - Thoracic medial branch blocks with bupivacaine and steroid
- Total: Total of all reporting groups
Arm/Group | Group I - With Local Anesthetics | Group II - With Bupivacaine and Steroid | Total
Number analyzed (Participants) | 50 | 50 | 100
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 47 | 50 | 97
  >=65 years | 3 | 0 | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.7 (11.7) | 42.8 (12.3) | 43.8 (12.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 32 | 63
  Male | 19 | 18 | 37

OUTCOME MEASURES:

1. Primary Outcome: Numeric Rating Scale
Description: Numeric rating scale represented 0 with no pain and 10 with the worst pain imaginable.
Time Frame: 2 years
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Group I Without Steroids: Thoracic Facet Joint Nerve Blocks with Local Anesthetic (0.25% Bupivacaine)
- Group II With Steroid: Thoracic Facet Joint Nerve Blocks with Local Anesthetic (0.25% Bupivacaine) and Steroids (0.15 mg of non-particulate betamethasone)
Arm/Group | Group I Without Steroids | Group II With Steroid
Number analyzed (Participants) | 50 | 50
units on a scale
  Baseline | 7.9 (0.9) | 7.8 (1.0)
  3 months | 3.1 (0.9) | 3.1 (0.7)
  6 months | 3.0 (0.9) | 3.2 (0.8)
  12 months | 3.2 (0.9) | 3.1 (1.0)
  18 months | 3.0 (1.0) | 3.1 (1.0)
  24 months | 3.1 (1.2) | 3.1 (1.0)
Statistical Analysis 1: Comparison: Group I Without Steroids vs Group II With Steroid; Test type: Superiority or Other; p = 0.964, ANOVA

2. Other Pre Specified Outcome: Opioid Intake
Description: Opioid intake(morphine equivalence mg)
Time Frame: 24 months
Measure: Mean (Standard Deviation); unit: mg/day
Groups:
- Group I - Without Steroids: Thoracic medial branch blocks with local anesthetics
- Group II - With Steroids: Thoracic medial branch blocks with bupivacaine and steroid
Arm/Group | Group I - Without Steroids | Group II - With Steroids
Number analyzed (Participants) | 50 | 50
mg/day
  Baseline | 48.0 (53.75) | 47.9 (48.6)
  3 months | 38.0 (44.2) | 40.3 (33.9)
  6 months | 38.2 (46.1) | 39.3 (34.8)
  12 months | 37.6 (38.4) | 37.8 (33.2)
  18 months | 37.6 (46.4) | 38.7 (35.2)
  24 months | 37.6 (46.4) | 38.7 (35.2)
Statistical Analysis 1: Comparison: Group I - Without Steroids vs Group II - With Steroids; Test type: Superiority or Other; p = 0.892, ANOVA

3. Primary Outcome: Oswestry Disability Index
Description: Oswestry Disability Index (ODI) - ODI score is ranged from 0 to 50. Total score is converted in to percent disability. ODI Scoring: 0% to 20% (minimal disability), 21%-40% (moderate disability), 41%-60% (severe disability), 61%-80% (crippled) and 81%-100 (these patients are either bed-bound or exaggerating their symptoms).
Time Frame: 24 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Group I - Without Steroids | Group II - With Steroids
Number analyzed (Participants) | 50 | 50
units on a scale
  Baseline | 27.1 (6.6) | 27.5 (5.8)
  3 months | 13.0 (4.9) | 11.6 (3.7)
  6 months | 13.0 (4.2) | 11.9 (3.8)
  12 months | 12.0 (4.0) | 11.8 (3.9)
  18 months | 12.0 (4.9) | 11.7 (3.9)
  24 months | 11.7 (4.9) | 11.0 (4.2)
Statistical Analysis 1: Comparison: Group I - Without Steroids vs Group II - With Steroids; Test type: Superiority or Other; p = 0.560, ANOVA

ADVERSE EVENTS:
Arm/Group | Group I - With Local Anesthetics | Group II - With Bupivacaine and Steroid
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/50
Other Adverse Events (participants affected / at risk) | 0/50 | 0/50

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No